CLINICAL TRIAL: NCT03652116
Title: Subrectal and Subcutaneous Wound Infiltration With Bupivacaine Versus Pethidine for Postcesarean Section Pain Relief: a Randomized Clinical Trial
Brief Title: Bupivacaine Verus Pethidine for Post Cesarean Section Pain Relief
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Safwat, Lecturer in Obstetrics and Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PostCSLA
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Obstetric Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to local infiltration of cesarean section wound with either bupivacaine or pethidine; with follow up of postoperative pain relief.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine Group (Active Comparator): Patients delivered by cesarean section followed by wound infiltration by bupivacaine.
  Interventions: Drug: Wound infiltration by Bupivacaine
- Pethidine Group (Active Comparator): Patients delivered by cesarean section followed by wound infiltration by pethidine.
  Interventions: Drug: Wound infiltration by Pethidine

INTERVENTIONS:
Drug: Wound infiltration by Bupivacaine — Subcutaneous and subrectal infiltration with 0.25 % Bupivacaine diluted in 20 ml normal saline before closure of the wound
  Arms: Bupivacaine Group
Drug: Wound infiltration by Pethidine — Subcutaneous and subrectal infiltration with 50 mg pethidine diluted in 20 ml normal saline before closure of the wound
  Arms: Pethidine Group

SUMMARY:
The aim of this study is to compare between the effect of wound infiltration with bupivacaine or pethidine for post cesarean section pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Mode of delivery: Cesarean section.
* Gestational age: 37-40 weeks.
* Type of anaesthesia: Spinal anaesthesia.
* No past history of any medical disorder or other medical complications during pregnancy.

Exclusion Criteria:

* Women with known hypersensitivity to bupivacaine or pethidine.
* Women delivered vaginally.
* Women delivered under general anaesthesia.
* Women with known neurological or psychological disease.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Postoperative wound pain: VAS | first 24 hours postoperatively
  Postoperative wound pain will be assessed using visual analogous scale (VAS) ranging from 0 (no pain) to 10 (worst pain imaginable). Mean values will be calculated and compared between the three groups

SECONDARY OUTCOMES:
Total dose of opioid drugs needed | first 24 hours postoperatively
  Total dose of extra opioid drugs needed to achieve postoperative analgesia
Incidence of nausea and vomiting | first 24 hours postoperatively
  Number of patients experiencing nausea and vomiting
Incidence of urine retention | first 24 hours postoperatively
  Number of patients experiencing urinary retention
Incidence of hypotension | first 24 hours postoperatively
  Number of patients experiencing hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Samy, MD, Study Director — M Samy
Locations (1):
- Ain SHams Maternity Hospital, Cairo, Abbaseya, Egypt